CLINICAL TRIAL: NCT02436707
Title: A Multi-Stage Randomized Phase II Study of Novel Combination Therapy in the Treatment of Relapsed and Refractory Aggressive B-Cell Lymphoma
Brief Title: Novel Combination Therapy in the Treatment of Relapsed and Refractory Aggressive B-Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Cancer Trials Group (Network)
Collaborators: Janssen, LP (Industry); Roche Pharma AG (Industry); Karyopharm Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LY17
Record Dates: First submitted 2015-05-04; First posted 2015-05-07 (Estimated); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Lymphoma
MeSH Terms: conditions — Lymphoma | interventions — ibrutinib; Rituximab; Gemcitabine; Dexamethasone; Cisplatin; Mesna; Cyclophosphamide; Etoposide; Granulocyte Colony-Stimulating Factor; selinexor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- R-GDP (Active Comparator): Rituximab - 375 mg/m2 IV, 1.5 - 6 hours D1 (prior to cisplatin);
  Gemcitabine - 1000 mg/m2, IV 30 min D1, D8;
  Dexamethasone - 40 mg daily PO D1 - D4;
  Cisplatin - 75 mg/m2 IV, 1 hour D1;
  Interventions: Drug: Rituximab; Drug: Gemcitabine; Drug: Dexamethasone; Drug: Cisplatin
- Ibrutinib plus R-GDP (ACCRUAL COMPLETE) (Experimental): Ibrutinib 560 mg PO -- D1 - D21
  Rituximab 375 mg/m2 IV 1.5 - 6 hours D1 (prior to cisplatin)
  Gemcitabine 1000 mg/m2 IV 30 min D1, D8
  Dexamethasone 40 mg daily PO -- D1 - D4
  Cisplatin 75 mg/m2 IV 1 hour D1
  Interventions: Drug: Ibrutinib; Drug: Rituximab; Drug: Gemcitabine; Drug: Dexamethasone; Drug: Cisplatin
- R-DICEP (ACCRUAL COMPLETE) (Experimental): Rituximab 375 mg/m2 IV 1.5-6hrs Day 1 and Day 5 prior to Cisplatin
  Mesna 1.75 g/m2 IV 24 hour Cycle 1, Day 2, Day 3 and Day 4
  Cyclophosphamide, 1.75 g/m2 IV 2 hours, Day 2, Day 3 and Day 4
  Etoposide 350 mg/m2 IV 2 hours, Day 2, Day 3 and Day 4
  Cisplatin 35 mg/m2 IV, 2 hours, Day 2, Day 3 and Day 4
  G-CSF 300 mcg (<60kg); 480 mcg (60-90kg); 600 mcg (>90kg); SC, Daily, starting Day 15 until apheresis completed.
  Interventions: Drug: Rituximab; Drug: Cisplatin; Drug: Mesna; Drug: Cyclophosphamide; Drug: Etoposide; Drug: G-CSF
- Selinexor + R-GDP (Experimental): Selinexor - 40mg PO, D1, D3, D8
  Rituximab - 375 mg/m2 IV, 1.5 - 6 hours D1 (prior to cisplatin);
  Gemcitabine - 1000 mg/m2, IV 30 min D1, D8;
  Dexamethasone - 40 mg daily PO D1 - D4;
  Cisplatin - 75 mg/m2 IV, 1 hour D1;
  Interventions: Drug: Rituximab; Drug: Gemcitabine; Drug: Dexamethasone; Drug: Cisplatin; Drug: Selinexor

INTERVENTIONS:
Drug: Ibrutinib
  Arms: Ibrutinib plus R-GDP (ACCRUAL COMPLETE)
Drug: Rituximab
Drug: Gemcitabine
  Arms: Ibrutinib plus R-GDP (ACCRUAL COMPLETE); R-GDP; Selinexor + R-GDP
Drug: Dexamethasone
  Arms: Ibrutinib plus R-GDP (ACCRUAL COMPLETE); R-GDP; Selinexor + R-GDP
Drug: Cisplatin
Drug: Mesna
  Arms: R-DICEP (ACCRUAL COMPLETE)
Drug: Cyclophosphamide
  Arms: R-DICEP (ACCRUAL COMPLETE)
Drug: Etoposide
  Arms: R-DICEP (ACCRUAL COMPLETE)
Drug: G-CSF
  Arms: R-DICEP (ACCRUAL COMPLETE)
Drug: Selinexor
  Arms: Selinexor + R-GDP

SUMMARY:
The purpose of this study is to find out what effects new combinations of treatment will have this disease. New promising treatment strategies will be added to this study as they are available to be compared against the standard treatment.

DETAILED DESCRIPTION:
This research is being done to try to find new combinations of treatment that may be better for treating patients with this disease. It is not clear however if these treatments can offer better results than standard treatment.

The study uses a "pick the winner" design to facilitate efficient screening of novel combination treatment regimens and select those meeting pre-specified criteria for testing in the phase III setting. All novel treatment options will be compared against the standard treatment for this disease: rituximab plus gemcitabine, dexemthasone, and cisplatin (R-GDP).

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologic diagnosis for one of the following histologies according to the World Health Organization: documented at initial diagnosis or at relapse:

  * Diffuse large cell lymphoma, B-cell (includes primary mediastinal B-cell lymphoma, T-cell rich B-cell lymphoma);
  * Previous indolent lymphoma (follicular lymphoma, marginal zone lymphoma, including extranodal MALT lymphoma, lymphoplasmacytoid lymphoma) with transformation to diffuse large B-cell lymphoma at most recent relapse (biopsy proof of transformation is mandatory);
  * Unclassifiable B-cell lymphoma with indeterminate features between diffuse large B-cell lymphoma and Burkitt lymphoma.
* Biopsy proof of disease at initial diagnosis is mandatory. A repeat biopsy in primary refractory disease is preferred but not mandatory to confirm progressive disease. A biopsy at relapse is preferred but not mandatory. Participating centres must designate a local reference expert pathologist who will confirm the diagnosis for the patients enrolled at that centre.
* Patients must be CD20+ in order to be eligible for the study.
* Clinically and/or radiologically measurable disease (one site bidimensionally measurable). Measurements/ evaluations must be done within 28 days prior to randomization.
* Prior FDG-PET scan, if done at baseline, must be positive (known FDG-avid lymphoma)
* Patients with de novo aggressive B-cell lymphoma must have relapsed or progressed, or have refractory disease, after 1 prior line of therapy (R-CHOP chemotherapy or equivalent). Patients with histological transformation from low grade lymphoma may have had up to 3 prior treatment regimens. Patients with transformed low grade lymphoma treated with a non-anthracycline regimen may be enrolled at investigator discretion.
* Patient age is ≥16 years. Patients older than 65 years of age are not recommended for this study.
* ECOG performance status of 0, 1 or 2.
* Patient must be considered fit for intensive chemotherapy and ASCT, and an appropriate candidate to receive second-line salvage chemotherapy and ASCT.
* Life expectancy > 90 days.
* Laboratory Requirements: (must be done within 14 days of randomization)

Hematology:

* Granulocytes (AGC) ≥ 1.0 x 10^9/L (independent of growth factor support)
* Platelets ≥ 100 x 10^9/L (50 x 10^9/L if bone marrow involvement by lymphoma, independent of transfusion support)

Biochemistry:

* AST and ALT ≤ 3x ULN (if both are done, both must be <3x UNL)
* Serum total bilirubin ≤ 1.5x ULN (≤ 5x ULN if Gilberts Disease)
* Serum Creatinine ≤ 1.5x ULN (or estimated GFR of ≥ 40 mL/min/1.73m2 using Cockcroft Gault formula).

Women must be post-menopausal, surgically sterile or use reliable forms of contraception while on study. Women of child bearing potential and men who are sexually active must be practicing a highly effective method of birth control during and after the study consistent with local regulations regarding the use of birth control methods for subjects participating in clinical trials. Men must agree to not donate sperm during and after the study. These restrictions apply for 12 months (1 year) after the last dose of study drug.

* Women of childbearing potential must have a pregnancy test taken (either by serum beta-human chorionic gonadotropin [B-hCG]) or urine) and proven negative within 14 days prior to randomization. Women who are pregnant or breastfeeding are ineligible for this study.

Patient consent must be appropriately obtained in accordance with applicable local and regulatory requirements. Each patient must sign a consent form prior to enrollment in the trial to document their willingness to participate.

Patients must be accessible for treatment and follow up. Patients randomized on this trial must be treated and followed at the participating centre. This implies there must be reasonable geographical limits (for example: 1 ½ hour's driving distance) placed on patients being considered for this trial. Investigators must assure themselves the patients randomized on this trial will be available for complete documentation of the treatment, response assessment, adverse events, and follow-up.

In accordance with CCTG policy, protocol treatment is to begin within 5 working days of patient randomization.

Exclusion Criteria:

* Patients with a history of other malignancies, except: adequately treated non-melanoma skin cancer and superficial bladder cancer, curatively treated in-situ cancer of the cervix or breast, or localized excised prostate cancer, other solid tumours curatively treated with no evidence of disease for ≥ 3 years.
* Active and uncontrolled central nervous system involvement, meningeal or parenchymal. Patients with CNS disease at initial presentation and who are in a CNS CR at the time of relapse are eligible. MRI scanning and / or lumbar puncture should be performed if there is clinical suspicion of active CNS disease.
* Major surgery performed within 10 days of randomization.
* Known history of human immunodeficiency virus (HIV), active Hepatitis C Virus infection, active Hepatitis B Virus infection or any uncontrolled active systemic infection requiring intravenous (IV) antibiotics. Patients with Hepatitis B serology suggestive of infection are eligible if they are HBV DNA negative and concurrently treated with anti-viral therapy. Patients with a past history of hepatitis C who have eradicated the virus are eligible.
* Patients who have been vaccinated with live, attenuated vaccines within 4 weeks of randomization.
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure, or myocardial infarction within 6 months of Screening, or any Class 3 (moderate) or Class 4 (severe) cardiac disease as defined by the New York Heart Association Functional Classification.
* Any serious active disease or co-morbid medical condition, including psychiatric illness, judged by the local investigator to preclude safe administration of the planned protocol treatment or required follow-up.
* Any other serious intercurrent illness, life threatening condition, organ system dysfunction, or medical condition judged by the local investigator to compromise the subject's safety, interfere with the absorption or metabolism of selinexor tablets, or preclude safe administration of the planned protocol treatment or required follow-up, including (for example):

  * active, uncontrolled bacterial, fungal, or viral infection;
  * clinically significant cardiac dysfunction or cardiovascular disease.
* Pregnant or lactating females, or women of childbearing potential not willing to use an adequate method of birth control for the duration of the study.
* Patients are not eligible if they have a known hypersensitivity to the study drugs or their components.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2015-10-27 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Measure overall response rate | 2 years
  To determine the overall response rate (complete and partial response) to novel combination therapy in patients with relapsed and refractory aggressive B cell lymphoma

SECONDARY OUTCOMES:
Number and severity of adverse events | 2 years
  To evaluate the tolerability and toxicity of novel combinations. Adverse events will be monitored on an ongoing basis by the central office and their frequencies reported annually at investigators' meetings. Safety and tolerability will be reviewed in the first six patients assigned to ibrutinib plus R-GDP as part of a safety run-in. Ibrutinib dose will be reduced for subjects subsequently enrolled if necessary
Transplantation rate | 2 years
  A non-inferiority analysis of transplantation rate will be conducted with 10% non-inferiority margin. The one-sided 80% asymptotic confidence limit of the difference in transplantation rate will be calculated between treatment and control arms.
Stem cell collection rate | 2 years
  Stem cell collection rate defined as collection of ≥ 2 x 106 CD34+ cells/kg.
Event free Survival Rate | 2 years
  • Event free survival (EFS) at one year defined as time from study entry to any treatment failure including disease progression, or discontinuation of treatment for any reason
Overall Survival | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Michael Crump, Study Chair — Univ. Health Network-OCI/Princess Margaret Hospital, Toronto ON Canada; John Kuruvilla, Study Chair — Univ. Health Network-Princess Margaret Hospital, Toronto ON Canada
Locations (11):
- Canada (11):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BCCA - Vancouver, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Ottawa Hospital Research Institute, Ottawa, Ontario
  - University Health Network, Toronto, Ontario
  - CHUM-Centre Hospitalier de l'Universite de Montreal, Montreal, Quebec
  - CHU de Quebec-Hopital l'Enfant-Jesus (HEJ), Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

IPD SHARING:
Plan to Share IPD: Yes
Subject to CCTG Policy
URL: https://www.ctg.queensu.ca/public/policies

REFERENCES:
- [Result] Stewart DA, Kuruvilla J, Lee D, Dudebout JJ, Chua N, Larouche JF, Baetz T, Shafey M, Abdel-Samad N, Robinson S, Fleury I, Fraser G, Skrabek P, Kukreti V, Kelly J, Hay AE, Shepherd LE, Chen BE, Crump M. Canadian cancer trials group LY.17: A randomized phase II study evaluating novel salvage therapy pre-autologous stem cell transplant in relapsed/refractory diffuse large B-cell lymphoma-outcome of rituximab-dose-intensive cyclophosphamide, etoposide, cisplatin (R-DICEP) versus R-GDP. Br J Haematol. 2024 Sep;205(3):881-890. doi: 10.1111/bjh.19555. Epub 2024 May 27. PMID 38802107